CLINICAL TRIAL: NCT02880059
Title: Incidence and Effects of Sleep Apnea on Intracerebral Aneurysms - IESA-Study
Brief Title: Incidence and Effects of Sleep Apnea on Intracerebral Aneurysms
Acronym: IESA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Sebastian Zaremba, Dr. med. Sebastian Zaremba, University Hospital, Bonn
Other Study IDs: IESA-Study
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Sleep Apnea (Defined as Apnea Hypopnea Index > 5/h); Intracranial Aneurysm Size; Blood Pressure Medication; Comorbidities; Complications (Subarachnoid Hemorrhage)
Keywords: Sleep Apnea, Aneurysm, Subarachnoid Hemorrhage, Blood Pressure.
MeSH Terms: conditions — Sleep Apnea Syndromes; Subarachnoid Hemorrhage; Aneurysm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Cardiorepiratory Polygraphy — Sleep apnea screening by out-of-center polysomnography/polygraphy
  Other Names: Sleep Apnea Screening

SUMMARY:
Patients with intracerebral aneurysm will be screened for sleep apnea using out of center polysomnography/polygraphy. Baseline blood pressure and medication will be assessed. Patients will be followed for up to 5 years to examine the increase in aneurysm size, rupture rate and changes in medication.

DETAILED DESCRIPTION:
Patient presenting to the outpatient center for neurological of neurosurgical management of intracerebral aneurysm will be recruited. Sleep apnea will be assessed by questionnaire and out of center polygraph/polysomnography. Medication, comorbidities and blood pressure will be recorded. Change in aneurysm size and blood pressure medication will be evaluated annually for up to 5 years. Frequency of subarachnoid hemorrhage and increase in aneurysm size will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Intracerebral aneurysm
* Age >= 18yrs.
* Ability to give informed consent

Exclusion Criteria:

* Stroke within 3 month of study inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18yrs. and older with intracerebral aneurysm.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Blood pressure medication | Baseline
  Blood pressure medication at baseline will be accessed.
Blood pressure | Baseline
  Blood pressure on baseline visit will be accessed.

SECONDARY OUTCOMES:
Subarachnoid hemorrhage | 5 years
  Rate of aneurysm rupture and subarachnoid hemorrhage will be accessed annually.
Increase in size of aneurysm | 5 years
Change in blood pressure medication | 5 years
  Blood pressure medication will be accessed on annual follow-up for up to 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Erdem Gueresir, MD, PhD, Principal Investigator — Vice Chair of Department of Neurosurgery; Sebastian Zaremba, MD, Principal Investigator — Staff Physician
Locations (1):
- Department of Neurology and Department of Neurosurgery, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zaremba S, Albus L, Hadjiathanasiou A, Vatter H, Wullner U, Guresir E. Aneurysm size and blood pressure severity in patients with intracranial aneurysms and sleep apnea. J Clin Sleep Med. 2022 Jun 1;18(6):1539-1545. doi: 10.5664/jcsm.9906. PMID 35088709